CLINICAL TRIAL: NCT04212975
Title: TMJ Lavage Followed by Dextrose Prolotherapy
Brief Title: Arthrocentesis Followed by Prolotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Atef Fouda, clinical professor, Cairo University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Cairo University-11022
Record Dates: First submitted 2019-12-15; First posted 2019-12-30 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: TMJ Pain
Keywords: tmj; pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Glucose

STUDY DESIGN:
Masking Description: assessment of improvement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group 1 (Experimental): lavage by dextrose
  Interventions: Other: joint lavage with dextrose

INTERVENTIONS:
Other: joint lavage with dextrose — joint lavage with dextrose

SUMMARY:
we will do tmj joint lavage and followed by dextrose injection

DETAILED DESCRIPTION:
Two groups of patients one group will receive lavage with saline and other group will receive lavage then dextrose injection

ELIGIBILITY:
Inclusion Criteria:

* tmj painful joints patients healthy patients disk displacement with reduction

Exclusion Criteria:

* patients previously treated males young age group

Ages: 19 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-08 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
pain scores | 3 months
  Change in pain symptoms measured by visual analogue scale 1=better-to-10 worse
Maximum mouth opening measured in millimeter 36mm=normal, less than 36mm=worse | 3 months
  Change in mouth opening- decrease =worse

SECONDARY OUTCOMES:
Change in pain symptoms measured by visual analogue scale | 3 months
  Measurement of change in pain scores from 1-10, 1=better-to-10 worse

CONTACTS AND LOCATIONS:
Overall Officials: Atef Abd El H Fouda, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No